CLINICAL TRIAL: NCT04059913
Title: A Prospective, Randomized, Open-Label, Multi-Center Study to Evaluate the Efficacy and Safety of Multiple Roxadustat Dosing Regimens for the Treatment of Anemia in Dialysis Subjects With Chronic Kidney Disease
Brief Title: Evaluate the Efficacy and Safety of Multiple Roxadustat Dosing Regimens for the Treatment of Anemia in Dialysis Participants With Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-818
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: CKD Anemia in Dialysis Participants
Keywords: Anemia; Chronic Kidney Disease Dialysis; hemoglobin; End stage renal disease
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: ESA-Naïve Participants - Low Weight Based Dosing (Experimental): ESA-naïve participants will receive roxadustat 70 mg TIW for body weight 45 to <60 kg or 100 mg TIW for body weight ≥60 kg.
  Interventions: Drug: Roxadustat
- Part 1: ESA-Naïve Participants - Standard Weight Based Dosing (Experimental): ESA naïve participants will receive roxadustat 100 mg TIW for body weight 45 to <60 kg or 120 mg TIW for body weight ≥60 kg.
  Interventions: Drug: Roxadustat
- Part 1: ESA-Treated Participants - Low Weight Based Dosing (Experimental): ESA-treated participants will receive roxadustat 70 mg TIW for body weight 45 to <60 kg or 100 mg TIW for body weight ≥60 kg.
  Interventions: Drug: Roxadustat
- Part 1: ESA-Treated Participants - Standard Weight Based Dosing (Experimental): ESA treated participants will receive roxadustat 100 mg TIW for body weight 45 to <60 kg or 120 mg TIW for body weight ≥60 kg.
  Interventions: Drug: Roxadustat
- Part 2: Roxadustat QW (Experimental): Participants will receive roxadustat once a week (QW). Roxadustat dose will be 2-dose step increase from originally planned week 21 TIW per dose amount.
  Interventions: Drug: Roxadustat
- Part 2: Roxadustat BIW (Experimental): Participants will receive roxadustat twice a week (BIW). Roxadustat dose will be 1-dose step increase from originally planned week 21 TIW per dose amount.
  Interventions: Drug: Roxadustat
- Part 2: Roxadustat TIW (Experimental): Participants will receive roxadustat TIW. Roxadustat dose will continue per dose adjustment guideline.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be dosed orally per dose and schedule specified in the arm description.
  Other Names: FG-4592

SUMMARY:
This is a randomized, open-label, multi-center study in dialysis chronic kidney disease (CKD) participants to evaluate the efficacy and relative safety of different dosing regimens of roxadustat over a 36-week treatment period.

There are 3 study periods:

* Screening Period (up to 4 weeks)
* Treatment Period (36 weeks)

Part 1: Correction/Conversion Period (Weeks 1-20)

Part 2: Hemoglobin (Hb) Maintenance Period (Weeks 21-36)

* Follow-up Period (4 weeks)

DETAILED DESCRIPTION:
Approximately 102 erythropoiesis stimulating agents (ESA)-naïve participants and 204 ESA-treated participants will be enrolled and randomized respectively in a 1:1 ratio to receive roxadustat at one of 2 starting doses as below:

* Low weight-based dosing: 70 milligrams (mg) 3 times a week (TIW) for body weight <60 kilograms (kg) or 100 mg TIW for body weight ≥60 kg
* Standard weight-based dosing: 100 mg TIW for body weight <60 kg or 120 mg TIW for body weight ≥60 kg

After 20 weeks of treatment, all eligible participants whose last 2 Hb levels ≥105 grams (g)/liter (L) and change in Hb over the most recent 4 weeks is > - 10 g/L will switch to receive roxadustat for another 16 weeks to evaluate the efficacy and safety of new dosing regimens.

At the end of Week 36, all participants will discontinue roxadustat and enter a 4-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. CKD with end-stage renal disease (ESRD) on either hemodialysis (HD) or peritoneal dialysis (PD)

Exclusion Criteria:

1. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibody (anti-HCV Ab).
2. Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thromboembolic event (for example, deep venous thrombosis or pulmonary embolism) within 26 weeks prior to Day 1.
3. History of malignancy, myelodysplastic syndrome, and multiple myeloma.
4. Chronic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (for example, systemic lupus erythematosis [SLE], rheumatoid arthritis, celiac disease).
5. Clinically significant gastrointestinal bleeding.
6. Women of childbearing potential and men with sexual partners of child bearing potential who are not using adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Part 1 (ESA Naïve): Percentage of Participants who Achieved Hb ≥110 g/L in the First 20 Weeks | Weeks 1 to 20
Part 1 (ESA Treated): Percentage of Participants who Achieved Mean Hb ≥100 g/L Averaged Over Weeks 17 to 21 Visits | Weeks 17 to 21
Part 2: Mean Hb Value Averaged Over Weeks 33 to 37 Visits | Weeks 33 to 37

SECONDARY OUTCOMES:
Part 1: Mean Change in Hb Level From Baseline to Average Over Weeks 17 to 21 Visits | Baseline, Weeks 17 to 21
Part 1 (ESA-Naïve): Percentage of Participants With Mean Hb (Averaged Weeks 17 to 21 Visits) ≥100 g/L | Weeks 17 to 21
Part 2: Percentage of Participants With Mean Hb (Averaged Weeks 33 to 37 Visits) ≥100 g/L | Weeks 33 to 37

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Investigational Site, Hefei, Anhui
  - Investigational Site, Lanzhou, Gansu
  - Investigational Site, Guangzhou, Guangdong
  - Investigational Site, Shenzhen, Guangdong
  - Investigational Site, Nanning, Guangxi
  - Investigational Site, Zhengzhou, Henan
  - Investigational Site, Wuhan, Hubei
  - Investigational Site, Changsha, Hunan
  - Investigational Site, Baotou, Inner Mongolia
  - Investigational Site, Nanjing, Jiangsu
  - Investigational Site, Nanchang, Jiangxi
  - Investigational Site, Changchun, Jilin
  - Investigational Site, Shenyang, Liaoning
  - Investigational Site, Taiyuan, Shanxi
  - Investigational Site, Xi’an, Shanxi
  - Investigational Site, Chengdu, Sichuan
  - Investigational Site, Hangzhou, Zhejiang
  - Investigational Site, Beijing
  - Investigational Site, Shanghai
  - Investigational Site, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278